CLINICAL TRIAL: NCT05725356
Title: Effectiveness of Physical Exercise on Job Stress and Quality of Life in Office Workers With Chronic Non-Specific Neck Pain: A Randomized Controlled Trial
Brief Title: Effectiveness of Physical Exercise on Chronic Non-Specific Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qassim University (Other)
Collaborators: University of Tabuk (Other)
Responsible Party: Principal Investigator, Sattam Almutairi, Assistant professor, Qassim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UT-153-31-2021
Record Dates: First submitted 2023-01-31; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Receiving physical exercise treatment (basic body awareness therapy and neck-specific training exercises) and ergonomic modification
  Interventions: Other: Basic body awareness therapy
- Control (Other): Receiving ergonomic modification only
  Interventions: Other: Basic body awareness therapy

INTERVENTIONS:
Other: Basic body awareness therapy — Participants were instructed to focus on maintaining good posture, balance, uninterrupted breathing, increased awareness, and decreasing unnecessary muscle tension.
  Other Names: ergonomic modification

SUMMARY:
Neck pain is a common medical condition among office workers all over the world. The purpose of this study was to see if physical exercise, such as basic body awareness, neck-specific training exercises, and ergonomic modifications, could help reduce pain, disability, and job stress while also improving quality of life among office workers. Participants will be assigned at random to either an experimental (exercise therapy and ergonomic modification) or a control group (ergonomic modification).

ELIGIBILITY:
Inclusion Criteria:

* Age 25-60 years
* Greater than 3 months of chronic NSNP.
* Office workers and computer users
* The ability to continue working

Exclusion Criteria:

* A history of severe injury
* Previous physical therapy treatments
* Joint instability
* Frequent migraines
* Spasmodic torticollis
* Inflammatory rheumatic diseases
* Peripheral nerve entrapment
* Severe psychiatric illness
* Pregnancy
* Other conditions that prevent physical loading.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | Change from baseline pain at 8 weeks
  Used to assess pain intensity. It uses the numbers from 0 to 10 and 0 indicates (no pain) through 1-3 (mild pain, slight impairment in daily life activities), 4-6 (moderate pain, substantial impairment in daily life activities), and 7-10 (severe pain, severe impairment in daily life activities).
Neck Disability Index | Change from baseline pain at 8 weeks
  Patient's self-reported impairment due to neck pain. It is a self-reported tool comprising 10 items. Each item is graded on a 6-point scale ranging from 0 (no disability) to 5 (severe disability).

SECONDARY OUTCOMES:
Health and Safety Executive Management Standards Indicator Tool | Change from baseline pain at 8 weeks
  Assessing psychosocial stress in the work area. Thirty-five HSE-MS questions measure seven dimensions, including demands, control, supervisory support , peer support , relationships, role (including a clear understanding of the employee's role in the organization), and changes. A higher score on each dimension (5 points) indicated lower stress.
The Short Form Health Survey | Change from baseline pain at 8 weeks
  Used to measure the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sattam M Almutairi, Principal Investigator — Physical Therapy Department, College of Medical Rehabilitation Sciences, Qassim University
Locations (1):
- King Fahad Specialist Hospital, Buraidah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No